CLINICAL TRIAL: NCT06406504
Title: A Realistic Experience in Improving Pressure Injury Classification and Assessment Skills: In Situ Simulation and Moulage
Brief Title: Improving Pressure Injury Classification and Assessment Skills: In Situ Simulation and Moulage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Hatice ERDEM ÖNDER, Dr., Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MehmetAkifU-SBF-HEÖ-01
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pressure Injury
Keywords: In-situ simulation; simulation-based training; moulage; pressure injury; nursing students
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned to in-laboratory simulation group, in-situ simulation group, and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in-laboratory simulation group (Experimental): The simulation practices of the students in the simulation practices of the students in the simulation in-laboratory simulation group (n=30) were performed with moulage application on a standardised patient in the simulation laboratory
  Interventions: Other: in-laboratory simulation group
- in-situ simulation group (Experimental): The simulation practices of the students in the simulation practices of the students in the in-situ simulation group (n=30) were performed with moulage application on a standardised patient in a clinic of a university hospital.
  Interventions: Other: in-situ simulation group

INTERVENTIONS:
Other: in-laboratory simulation group — The students in-laboratory group performed the simulation applications in the patient room in the simulation laboratory. One of the Stage 2 and one of the Stage 3 PI was created by the researcher with moulage to the heel and lateral malleolus area of the standardised patient taken to the patient room.
  Arms: in-laboratory simulation group
Other: in-situ simulation group — Students in the in-situ simulation group performed the simulation practices in a patient room in a clinic at a university hospital. One of the Stage 2 and one of the Stage 3 PI was created by the researcher with moulage to the heel and lateral malleolus area of the standardised patient taken to the patient room.
  Arms: in-situ simulation group

SUMMARY:
The aim of this study was to evaluate the effectiveness of in-situ simulation and moulage to improve nursing students' pressure injury classification and assessment skills. A randomized controlled model with a pretest-posttest control group was used in this study. The population of the study consists of a faculty of nursing at a state university. The sample consisted of 84 nursing students. The control group received simulation-based training using a pressure injury simulator on a standardised patient in the simulation laboratory, the in-laboratory simulation group received simulation-based training using moulage on a standardised patient in the simulation laboratory, and the in-situ simulation group received simulation-based training using moulage on a standardised patient in the clinic of a university hospital. The research data were collected by Descriptive Characteristics Form, Pressure Injury Knowledge Test, Pressure Injury Assessment Form, Performance Checklist, Students' Satisfaction and Self-Confidence Scale and Student Feedback Form.

DETAILED DESCRIPTION:
In this study, the reality of the environment was increased with the in-site simulation method, the physical reality was increased by ensuring that the standardised patient characteristics match with the patient characteristics in the real world with moulage, and the functional reality was increased by performing a wound classification and evaluation similar to the real wound with moulage. In this context, this study was conducted to determine the effect of in-situ simulation and moulage application in order to improve nursing students' skills in Pressure Injury (PI) classification and assessment.

For this purpose, there are three hypotheses guiding the research:

There will be a difference between the PI knowledge test scores of the groups. There will be a difference between the groups' ability to classification and assessment PI.

There will be a difference between the satisfaction and self-confidence levels of the groups.

This study was structured as a randomized, controlled experimental investigation with pretest and posttest control groups. It was conducted to evaluate the effectiveness of in situ simulation and moulage to improve nursing students' PI classification and evaluation skills. It was conducted at a nursing school in Turkey between September 2021 and May 2023. Simulation-based experiences were designed based on the INACSL Healthcare Simulation Standards of Best PracticeTM Simulation Design. The study design was reported following the guidelines of the Consolidated Standards of Reporting Trials (CONSORT).

The study population comprised senior nursing students (N=284). The sample size was calculated on the basis of previous studies evaluating the effectiveness of the moulage method in PI assessment skills. Based on the power analysis, the study's sample size was determined to be 84 (ɑ=0.10, 1-β=0.95) with 95% power and ɑ=0.10 error (90% confidence interval). Taking into account possible losses during the study, 90 students were included. Senior nursing students who had not previously performed classification and assessment of PI, who had not attended any course related to PI, and who volunteered to participate were included in the study. In order to ensure homogeneous distribution of students in terms of academic achievement score, a statistician who was not involved in the study randomised the students according to their grade point averages at the end of the third year using a website. The simulation practices of the students in the control group (n=30) were performed with a PI simulator on a standardised patient in the simulation laboratory, the simulation practices of the students in the simulation in-laboratory group (n=30) were performed with moulage application on a standardised patient in the simulation laboratory, and the simulation practices of the students in the in-situ simulation group (n=30) were performed with moulage application on a standardised patient in a clinic of a university hospital. Since two students from each of the three groups left the study, the study was completed with 84 students.

ELIGIBILITY:
Inclusion Criteria:

* Senior nursing students
* Nursing students who had not previously performed classification and assessment of PI
* Nursing students who volunteered to participate were included in the study

Exclusion Criteria:

* Nursing students who had previously performed classification and assessment of PI
* Nursing students who do not attend simulation training

Ages: 22 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Pressure Injury Skill | four week
  This form was prepared by the researcher based on the literature. The form consists of twenty-five items and the stages of the PI assessment. The student's performance was scored as "correctly applied" (2 points), "partially applied" (1 point), "not applied" and "incorrectly applied" (0 points). The student can get a maximum score of 50 and a minimum score of 0. The form was evaluated by the same experts.

SECONDARY OUTCOMES:
Pressure Injury Knowledge | four week
  The questionnaire was prepared by the researcher based on the literature. The PI knowledge test consists of 15 multiple-choice questions on PI general knowledge (5 questions), classification (7 questions) and PI assessment (3 questions). The highest score is 100 and the lowest score is 0. For the test, expert opinion was obtained from four faculty members, two of whom were faculty members working in the field of PI.
Students' satisfaction and self-confidence scale | four week
  This scale is used to measure students' satisfaction and self-confidence in a simulation learning environment. It comprises two sub-dimensions: "Satisfaction with Current Learning" and "Self-confidence in Learning." Student responses for each item were recorded on a five-point Likert-type scale; Strongly Disagree, Disagree, Neutral, Agree and Strongly Agree. It was found that the Cronbach's Alpha value for "Satisfaction with current learning" was 0.85 and Cronbach's Alpha value for "Self-confidence in Learning" was 0.77. Scores range from 1 to 5; 1 is the lowest score and 5 points is the highest and as the total score increases, students' satisfaction and selfconfidence in learning increase, as well.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice ERDEM ONDER, Principal Investigator — Mehmet Akif Ersoy University; Dilek SARI, Study Director — Ege University
Locations (1):
- Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

REFERENCES:
- [Derived] Erdem Onder H, Sari D. Improving pressure injury assessment skills of nursing students' using in-situ simulation and moulage: a randomized controlled trial. BMC Nurs. 2025 Nov 6;24(1):1373. doi: 10.1186/s12912-025-04049-x. PMID 41199277